CLINICAL TRIAL: NCT02883387
Title: CT-Angiography Prior to DIEP Flap Breast Reconstruction a Randomized Controlled Trial
Brief Title: CT-Angiography Prior to DIEP Flap Breast Reconstruction
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Colorado, Denver (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 15-2448
Record Dates: First submitted 2016-08-25; First posted 2016-08-30 (Estimated); Last update posted 2022-02-24 (Actual); Status verified 2022-02

CONDITIONS: Breast Cancer
Keywords: DIEP flap; Deep inferior epigastric artery perforator flap
MeSH Terms: conditions — Breast Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Preoperative CT Angiography (Experimental): Patients will receive preoperative CT angiography to map the blood vessels potentially used for reconstruction
  Interventions: Other: Preoperative CT angiography
- No Imaging Preoperatively (Active Comparator): No preoperative vessel mapping will be done
  Interventions: Other: No Preoperative Imaging

INTERVENTIONS:
Other: Preoperative CT angiography — Patients will receive a CT scan to map the blood vessels to be used during surgery for breast reconstruction
  Arms: Preoperative CT Angiography
Other: No Preoperative Imaging — No imaging will be done to map blood vessels prior to surgery
  Arms: No Imaging Preoperatively

SUMMARY:
This study will Investigate whether or not preoperative computed tomography (CT) angiography will lower operative times and post operative complications for breast reconstruction performed with a deep inferior epigastric artery perforator flap (DIEP).

ELIGIBILITY:
Inclusion Criteria:

* Planning breast reconstruction with DIEP flap
* Age 18 to 75 years

Exclusion Criteria:

* Mild to moderate loss of kidney function (Estimated Glomerular Filtration Rate (eGFR) < 60)
* Decisionally challenged
* Pregnant
* Hepatic failure

Ages: 18 Years to 75 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 39 (Actual)
Dates: Start 2016-09; Primary Completion 2020-03-01 (Actual); Study Completion 2020-03-01 (Actual)

PRIMARY OUTCOMES:
Total Operative Time | Time of incision to incision closure
  Time required to perform breast reconstruction with DIEP flap

CONTACTS AND LOCATIONS:
Overall Officials: David W Mathes, MD, Principal Investigator — University of Colorado, Denver
Locations (1):
- University of Colorado Anschutz Medical Campus, Aurora, Colorado, United States

IPD SHARING:
Plan to Share IPD: No